CLINICAL TRIAL: NCT00611182
Title: Dyspnea in Patients With Pulmonary Fibrosis
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: University of Chicago (Other); American College of Chest Physicians (Other); The John A. Hartford Foundation (Other); Association of Specialty Physicians, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: H5476-31357-01
Record Dates: First submitted 2008-01-28; First posted 2008-02-08 (Estimated); Last update posted 2013-11-18 (Estimated); Status verified 2013-11

CONDITIONS: Pulmonary Fibrosis
Keywords: dyspnea; pulmonary fibrosis; interstitial lung disease; shortness of breath
MeSH Terms: conditions — Pulmonary Fibrosis; Dyspnea; Lung Diseases, Interstitial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients with Pulmonary Fibrosis

SUMMARY:
This study has two aims:

1. To determine the relationship of shortness of breath (dyspnea) to other conditions present in patients with pulmonary fibrosis.
2. To define the relationship between shortness of breath and rate of functional decline in patients with pulmonary fibrosis.

DETAILED DESCRIPTION:
Idiopathic Pulmonary Fibrosis is the most common form of chronic fibrosing lung disease seen by pulmonologists, with an estimated 128,000 cases in the United States alone. It is almost surely a disorder related to aging, with a median age at the time of diagnosis of approximately 65 years; IPF is almost unheard of under the age of 50. Dyspnea is common in patients with IPF, and is often the primary symptom of the disease. It is tightly linked to quality of life in IPF, suggesting that the experience of dyspnea has wide-ranging and clinically-significant consequences. Despite its importance, surprisingly little is known about the etiology or functional impact of dyspnea in this disease.

This research proposal focuses on defining the relationship of dyspnea to comorbidity and the rate of functional decline in patients with IPF

Aim 1: To determine the relationship of dyspnea to other conditions present in patients with IPF.

Dyspnea is a complex symptom, related to both mechanical and cognitive factors. The mechanisms of dyspnea in IPF remain unknown, but there are several likely contributors that are both IPF and non-IPF related. Although IPF is a chronic disease of the elderly, no one has investigated the relationship between common geriatric conditions and dyspnea. It is well established that the perception of dyspnea depends equally on factors that influence the intensity of the experience of breathlessness (such as thoracic restriction and weakness) and the distress which that intensity produces. Gender, ethnicity, anxiety, pain, and depression all may contribute to the distress caused by dyspnea (and therefore its intensity) in IPF.

Aim 2: To define the relationship between dyspnea and rate of functional decline in IPF.

Numerous studies have looked at predictors of survival in patients with IPF, and both baseline and change in dyspnea over time have been shown to be significantly associated. The prediction of future morbidity, however, is largely unstudied. Established markers of functional decline in geriatric patients include weight loss, decline in walking speed over 4 meters, and the onset of disability as defined by the ability to perform activities of daily living (ADLs) and instrumental activities of daily living (IADLs). Dyspnea likely impacts patients' activity levels and/or motivation to stay active, and may contribute to worsening functional decline.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older with pulmonary fibrosis, and able to travel to University of California San Francisco for study visits

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: community sample
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2008-01; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Dyspnea | 6 months

SECONDARY OUTCOMES:
Functional status | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Harold R. Collard, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

REFERENCES:
- See also: UCSF Interstitial Lung Disease Program — http://www.ucsfhealth.org/ild